CLINICAL TRIAL: NCT00647569
Title: Randomized Controlled Trial of Collagen Mesh for Prevention of Ventral Hernia in Patients With Vertical Rectus Abdominis Musculocutaneus Flap for Advanced Pelvic Malignancy
Brief Title: Trial of Collagen Mesh for Prevention of Ventral Hernia After Surgery for Advanced Pelvic Cancer
Acronym: VRAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Cook Biotech Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VRAM M-20070240
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Incisional Hernia; Pelvic Cancer
Keywords: vertical rectus abdominis musculocutaneus flap; mesh repair; salvage surgery
MeSH Terms: conditions — Incisional Hernia; Pelvic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): No previous major abdominal surgery
  Interventions: Procedure: Mesh repair; Procedure: Conventional facial closure
- B (Experimental): Previous major abdominal surgery
  Interventions: Procedure: Mesh repair; Procedure: Conventional facial closure

INTERVENTIONS:
Procedure: Mesh repair — A Surgisis Gold Hernia repair graft (Cook Biotech Incorporated, West Lafayette, IN, U.S.A) is placed at the donor site of the rectus abdominis muscles used for the rotation flap before the abdominal fascia is sutured with continuous running suture.
  Other Names: Surgisis Gold Hernia repair graft
Procedure: Conventional facial closure — The abdominal facia is closed with with continuous running suture

SUMMARY:
The aim of the present project is to investigate whether use of biological mesh at the donor site of the rotation flap in closure of the abdominal wall reduce the frequency of incisional hernia formation compared to the usual abdominal wall closure after abdominal rotation flap operation in surgery for advanced pelvic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated with a vertical rectus abdominis musculocutaneus flap after abdominoperineal resection for advanced pelvic cancer.

Exclusion Criteria:

* Pre or perioperative knowledge of disseminated malignancy
* Unable to follow the control program
* Known allergy to pig
* Compromised immune defense
* Artificial heart valve or recent (< 3 months) implanted foreign body
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
incisional hernia formation determined by CT scan 1 year postoperative | 1 year postoperative

SECONDARY OUTCOMES:
postoperative morbidity | 30 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Peter Christensen, M.D., Ph.d, Principal Investigator — Department of Surgery P, Aarhus University Hospital, Denmark
Locations (1):
- Surgical Research Unit, Department of Surgery P, Aarhus University Hospital, Aarhus, Denmark